CLINICAL TRIAL: NCT06255483
Title: Anatomical Research of the Clavicular Pedicled Flap for Mandibular Reconstruction: Vascularization and Harvesting Technique
Brief Title: Anatomical Research of the Clavicular Pedicled Flap for Mandibular Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Tahar Maamouri University Hospital (Other)
Responsible Party: Principal Investigator, Imen Turki Mehri, MD, Principal investigator, Mohamed Tahar Maamouri University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Teaching Hospital Maamouri
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Mandibular Reconstruction; Maxillofacial Injuries
Keywords: Clavicle; Pedicled Flap; Bosniak Node; Microvascular Network; Mandibular reconstruction
MeSH Terms: conditions — Maxillofacial Injuries | interventions — Mandibular Reconstruction

STUDY DESIGN:
Intervention Model Description: The harvest of a pedicle osteoperiosteal clavicular flap was performed in the same way on ten fresh cadaveric specimens. The vascular supply was studied by colored latex and methylene blue injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteoperiosteal clavicular flap (Other): Harvesting of a pedicled osteoperiosteal clavicular flap and clarification of its vascular supply
  Interventions: Other: Osteoperiosteal pedicled clavicular flap for mandibular and facial bone reconstruction

INTERVENTIONS:
Other: Osteoperiosteal pedicled clavicular flap for mandibular and facial bone reconstruction — A clavicular flap with a vascular supply based on the transverse cervical artery which receives a reverse blood supply from the ascending cervical artery. This vascular pattern is reliable because of the existence of the sub-occipital microvascular network named the " Bosniak node ".
  Other Names: Anatomical Research of the clavicular pedicled flap for mandibular reconstruction

SUMMARY:
Because of the proximity of the clavicular bone to the oral cavity, and the suitable characteristics of the bone for implant placement, its use as a pedicled flap is an attractive method of mandibular reconstruction. This research, performed on fresh cadaver specimens, describes the vascular supply and harvesting technique of a pedicled clavicular bone allowing a mandibular reconstruction with a single surgical field.

DETAILED DESCRIPTION:
An osteoperiosteal clavicular flap was harvested from the right side, on 10 fresh male cadaver specimens whose age of death ranged between 42 and 65 years. The dissection was carried out by the investigator at the laboratory of the Anatomy of René Descartes University of Medicine in Paris in 2004, as well as in the Forensic Medicine Department of Mohamed Tahar Maamouri University Hospital in Tunisia.

Technical steps for harvesting the pedicled osteoperiosteal clavicular flap:

The cadaver is placed in dorsal recumbency, and a pad under the shoulders. A cervical incision with a " Z " shape was performed in which the upper branch was placed two centimeters below and parallel to the inferior jawline to preserve the marginal mandibular nerve. The vertical branch of the incision continued following the path of the sternocleidomastoid muscle and reached the lower branch of the " Z " at the level of the clavicle.

The dissection was carried out in the cervical region's sub-platysmal plane and the pre-pectoral and pre-deltoid planes. The deep plane can be approached through an incision of the superficial cervical fascia overlying the sternocleidomastoid muscle taking into consideration the spinal accessory nerve. Then, the clavicle was released from the sternocleidomastoid muscle, but the subclavius muscle insertion was preserved on the clavicle to protect the subclavian vein branches. The level of undermining dissection was confined to the loose fat pad overlaying the scalene muscle, within which the vessels are embedded without exposing the brachial plexus.

The anterior surface of the subclavian vein was exposed, and the vessels arising from this vein were ligated. The clavicular bone attached to a celluloadipous pedicle has been lifted exposing the thyrocervical trunk. A celluloadipous tissue around the branches of this trunk (cervical transverse artery, inferior thyroid artery, ascending cervical artery, and suprascapular artery) was preserved in their dissection, and care was taken to avoid injury of the phrenic nerve, noticeable near the inferior thyroid artery. Then, the cervical transverse and suprascapular arteries were ligated at their distal part. Nevertheless, the inferior thyroid artery could be also ligated, which increases the total pedicle length of the flap and improves its arc of rotation. Otherwise, the flap will be bi-pedicled. The ascending cervical artery was dissected along the anterior scalene muscle up to the level of the transverse process of the fourth cervical vertebrae which is considered the vascular pedicle rotation point.

The vascular supply of the clavicular flap was highlighted by injecting the thyrocervical trunk with coloured latex after ligating the following arteries at their distal parts: the inferior thyroid, the suprascapular, and the cervical transverse.

ELIGIBILITY:
Inclusion Criteria:

* Fresh cadaveric speciemen

Exclusion Criteria:

* Neck injury or previous neck dissection

Ages: 42 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Vasculature of the flap | Immediately after harvesting the flap
  Clavicular periosteal vessels emerging from the cervical transverse artery were highlighted and further identified after methylene blue injection
Facial accessibility | Immediately after harvesting the flap
  Mandibular and zygomatic region were reached by this flap
Bone characteristics | Immediately after harvesting the flap
  full-thickness bone with a length ranging between 9 and 11 centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Mohamed Tahar Maamouri, Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
This research has been published.
Supporting Information: CSR
Time Frame: Anatomical research of the clavicular pedicled flap for mandibular reconstruction: vascularization and harvesting technique
URL: https://link.springer.com/article/10.1007/s10006-023-01192-0